CLINICAL TRIAL: NCT04871828
Title: The Efficacy of Leukotriene Inhibitor in Adult Patients With Moderate SARS-COV-2 Symptoms (COVID19): (Randomized Clinical Trial)
Brief Title: The Efficacy of Leukotriene Inhibitor in Adult Patients With Moderate SARS-COV-2 Symptoms (COVID19)
Acronym: PROMISE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC20/206/R
Record Dates: First submitted 2021-05-01; First posted 2021-05-04 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Moderate Covid19
MeSH Terms: interventions — Leukotriene Antagonists

STUDY DESIGN:
Intervention Model Description: Prospective randomized placebo-controlled double-blinded clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Zafirlukast plus the standard treatment according to Saudi CDC protocol (combination experimental arm)
  Description of investigational drug Zafirlukast is leukotriene receptor antagonist (LTRA) for the maintenance treatment of asthma. It is available as a tablet and is usually dosed twice daily. It is approved by USFDA and currently commercially marketed under the name of Accolate 20 mg oral tablet. The drug will be acquired from the pharmacy and will be received by the patient during the hospital admission via research coordinator. The study drug will be stored in at room temperature (15 - 25 c) in the hospital's pharmacy and a delegated pharmacist will be responsible for dispensing and return of any drugs.
  The study drug will be administrated to the patient in the dose of 20 mg orally twice daily for 10 days (fixed dose with no staring or escalating dose).
  Interventions: Drug: Leukotriene Receptor Antagonist
- Control (Placebo Comparator): placebo plus the standard treatment according to Saudi CDC protocol
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Leukotriene Receptor Antagonist — Zafirlukast
  Arms: Treatment
Other: Placebo — Placebo
  Arms: Control

SUMMARY:
There is an urgent need to explore therapeutic options for SARS-CoV-2 in order to face the pandemic. The selected intervention was based on that zafirlukast will have dual effect; first it will block the virus replication through inhibiting the COVID19 helicase that is involved in virus replication and secondly by reducing the inflammation through antagonizing the leukotriene receptor.

The purpose of this study is to evaluate the clinical efficacy and safety of Leukotriene receptor antagonist in the treatment of moderate cases of COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or above
2. Diagnosed with COVID-19 by PCR confirmed SARS-coV-2 viral infection.
3. Able to sign the consent form and agree to clinical samples collection
4. Moderate symptomatic COVID-19 patients, (any or all of the followings: fever or cough or SOB)
5. Admitted to the hospital (outside the ICU)
6. Patients had to be enrolled within 10 days of symptoms onset.
7. willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

1. Asthmatic patient using antiasthma medications
2. Being in the hospital or in home isolation for more than 72 hours before the start of the study drug.
3. Known sensitivity/allergy to the study drug
4. Pregnancy
5. Patient refused
6. Chronic liver disease
7. Severe mental disorder
8. Unstable patients requiring ICU admission
9. Participating in other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-02-28 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement, | 28Day
  The time from symptoms resolved: No fever for 72 hours, no cough, no SOB or live discharge from the hospital, whichever came first.

SECONDARY OUTCOMES:
Escalate therapy. | 28Day
  The requirement to escalate therapy.
PCR test | Day14
  PCR test negative conversion rate at day 14
Length of hospital stay. | 28Day
  Length of hospital stay.
Duration of fever | 28Day
  Duration of fever

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz Medical city, MNGHA, Riyadh, Saudi Arabia